CLINICAL TRIAL: NCT01574963
Title: Graz Osteoprotegerin as a Risk Factor (GORF) Study: THE ROLE of OSTEOPROTEGERIN (OPG) and the RECEPTOR ACTIVATOR OF NUCLEAR FACTOR-Kb LIGAND (RANKL) IN PATIENTS REQUIRING SURGERY FOR CORONARY HEART DISEASE
Brief Title: Graz Osteoprotegerin as a Risk Factor (GORF) Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daniela Malliga, MD, OA Dr. med. univ., Medical University of Graz
Other Study IDs: GORF 2.0
Record Dates: First submitted 2012-04-04; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Prevalent OPG and RANKL Excession in Patients With CAD
Keywords: Coronary artery disease; OPG; RANKL; bone disease
MeSH Terms: conditions — Coronary Artery Disease; Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CAD Patients: Patients suffering from CAD requiring coronary artery bypass grafting
- Control Patients: Patients without CAD

SUMMARY:
Osteoprotegerin (OPG) is membrane bound in the immune system but can also be produced and secreted almost everywhere in the organism, so that it is mainly available in soluble form. So far, the OPG/RANKL/RANK system has been most intensively studied in bone. The binding of RANKL on its receptor RANK, which is expressed by osteoclasts, activates a number of osteoclastic cell functions. OPG also has a key function in the vascular system. Patients with coronary heart disease (CAD) have elevated OPG serum levels, probably as a sign of ischemic or inflammatory endothelial damage. Elevated OPG levels were also found in patients with advanced heart failure, whereby OPG correlated with pro BNP (brain natriuretic peptide) and was a predictor for cardiovascular morbidity and mortality.

Our prospective cohort study will include 150 men (75 patients requiring surgery for CAD and a control group without coronary heart disease). The primary endpoints are the differences between the two groups in serum levels of OPG and RANKL, markers of bone metabolism (osteocalcin [OC], crosslaps [CTX], tartrate resistant acid phosphatase (TRAP5b), 25(OH) vitamin D [Vit D], 1.25(OH) vitamin D, parathormone [iPTH], endocrine parameters related to vascular damage (e.g. aldosterone, renin and cortisol) and bone mineral density. Metabolomic based biomarkers will be evaluated to explore the mechanisms behind OPG-RANKL linked CVD damage. In the patients further studies of the mRNA expression of OPG, RANKL, TRAP5b, arginine:glycine amidinotransferase (AGAT) and osteocalcin in bone (sternum sliver) and vascular wall (aorta, internal thoracic artery and the great saphenous vein) will be performed.

A further study endpoint is the analysis of a causal coincidence between osteoporosis and CAD and the discrimination of possible key factors in the two entities. These will be determined by the correlation between the above-mentioned markers in serum and the expression in different vessels and in bone tissue.

In addition to analysis of the degree of vascular sclerosis, the mineral content of the bone will also be analyzed in a subpopulation with quantitative backscattered electron imaging (qBEI) related to the degree of vascular sclerosis and bone mineral density. The ultimate goal of the analysis is the discrimination of the most sensitive predictive marker(s) for diagnosis and outcome of patients with CAD for the purpose of early diagnosis and primary prevention of the disease.

CAD and osteoporosis are increasingly prevalent diseases that overlap. In both entities, OPG plays a role not only in pathogenesis but also as an outcome predictor. We aim to study the relevance of OPG concentration in serum but also in the vessel wall and the bone.

ELIGIBILITY:
Inclusion Criteria:

* Male patients above 40 years of age presenting with symptomatic CAD and scheduled for a coronary artery bypass graft (CABG) are eligible for the study. The control group includes male patients scheduled for elective surgery other than cardiac procedures.

Exclusion Criteria:

* Exclusion criteria are a second indication for heart surgery, chronic renal disease with a glomerular filtration rate < 30ml/min, advanced liver disease (AST, ALT, GGT > 3fold upper limit of normal), history of malignancy within the last 5 years and ongoing osteoprotective treatment.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients above 40 years of age presenting with symptomatic CAD and scheduled for a coronary artery bypass graft (CABG) are eligible for the study. The control group includes male patients scheduled for elective surgery other than cardiac procedures.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
OSTEOPROTEGERIN (OPG) | Baseline at time 0 (at the beginning of the study). The participants will be followed for the duration of hospital stay, an expected average of 10 days.
  The primary endpoints are the differences between the two groups in serum levels of OPG and RANKL, markers of bone metabolism (osteocalcin [OC], crosslaps [CTX], tartrate resistant acid phosphatase (TRAP5b), 25(OH) vitamin D [Vit D], 1.25(OH) vitamin D, parathormone [iPTH], endocrine parameters related to vascular damage (e.g. aldosterone, renin and cortisol) and bone mineral density.

SECONDARY OUTCOMES:
RANKL | At baseline. The participants will be followed for the duration of hospital stay, an expected average of 10 days.
  The primary endpoints are the differences between the two groups in serum levels of OPG and RANKL, markers of bone metabolism (osteocalcin [OC], crosslaps [CTX], tartrate resistant acid phosphatase (TRAP5b), 25(OH) vitamin D [Vit D], 1.25(OH) vitamin D, parathormone [iPTH], endocrine parameters related to vascular damage (e.g. aldosterone, renin and cortisol) and bone mineral density.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Malliga, MD, Principal Investigator — Medical University of Graz, Department of Surgery, Division for Cardiac Surgery; Astrid Fahrleitner-Pammer, Prof., Study Director — Medical University of Graz, Department of Internal Medicine, Division for Endocrinology and Metabolism; Doris Wagner, MD, Study Chair — Medical University of Graz, Department of Surgery, Division for Transplantation
Locations (1):
- Medical University of Graz, Graz, Austria